CLINICAL TRIAL: NCT00273988
Title: A Pharmacokinetic Study to Evaluate the Interaction Between Nevirapine (Viramune®) and Methadone in HIV-1 Infected, Opioid-dependent Adults on Stable Methadone Maintenance Therapy
Brief Title: Pharmacokinetic Study of Interaction Between Nevirapine and Methadone in HIV-1 Infected, Opioid-dependent Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1390
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Nevirapine

INTERVENTIONS:
Drug: nevirapine

SUMMARY:
The purpose of this study was to determine the effects of nevirapine treatment on the pharmacokinetics of methadone in HIV-1 infected, opioid-dependent adults who had been on a stable methadone maintenance therapy for at least five days prior to study entry.

DETAILED DESCRIPTION:
Ten HIV-1 infected, opioid-dependent adults on stable methadone treatment were to be enrolled in this study. This was an open-label, sequential treatment study, with methadone pharmacokinetics sampling before and after twenty-one (21) days of nevirapine administration.

All patients received the same regimen. Methadone was administered in the first treatment period, and combination treatment of methadone and nevirapine was given in the second treatment period. In the first period, patients received methadone at their current steady state dose. In the second period (study days 1-21), they also received nevirapine 200mg qd (study days 1 to 14) and 200mg bid (study days 15 to 21). Blood samples were taken at the start of the first treatment period and at the end of the second treatment period for analysis of methadone and nevirapine pharmacokinetics parameters.

Study Hypothesis:

It was expected that nevirapine would decrease methadone levels in this patient population.

Comparison(s):

The study compared methadone steady state exposure in the absence and presence of steady state nevirapine. A range of pharmacokinetics parameters were assessed including clearance of methadone (the primary endpoint variable), area under the concentration-time curve, maximum concentration, time to maximum concentration and minimum concentration (measured for both methadone and nevirapine).

ELIGIBILITY:
Inclusion criteria:

* Treatment-naïve, fulfilling standard criteria to commence antiretroviral therapy. Previous exposure to less than two weeks of nucleoside reverse transcriptase therapy was permitted. (Later amended to allow previous exposure to non-nucleoside reverse transcriptase inhibitor therapy (NNRTI) if the patient was off NNRTI therapy for at least two weeks prior to entry.)
* Plasma HIV-1 ribonucleic acid (RNA) assay performed at screening documenting HIV-1 infection or previous laboratory documentation of HIV-1 positive status.

CD4+ cell count at least 100 cells/mm3 (later amended to at least 50 cells/mm3), within 28 days prior to study day 0.

* Patients who met the following laboratory parameters:

  * Lymphocyte count at least 1 x 109/L
  * Haemoglobin at least 5.7 mmol/L [9.0 g/dL] (men and women)
  * Platelet count at least 75 x 109/L
  * Alkaline phosphatase less than or equal to 3 times the upper limit of normal
  * Serum glutamate oxaloacetate transferase (SGOT) and serum pyruvate oxaloacetate transferase (SGPT) less than or equal to 3 times the upper limit of normal
  * Total bilirubin less than or equal to 1.5 times the upper limit of normal
  * Serum creatinine less than or equal to 2.0 mg/dL.
* On stable methadone maintenance therapy for at least five days prior to entry.
* Patients of reproductive potential must have been willing to use a reliable method of double-barrier contraception (such as a diaphragm with spermicidal cream or jelly, or condoms with spermicidal foam).
* Informed of, and willing and able to comply with the investigational nature of the study, and have signed a written consent in accordance with ethics committee and regulatory guidelines.

Exclusion criteria:

* Female patients who were pregnant or breast-feeding.
* Systemic treatment with corticosteroids or drugs known to be hepatic enzyme inducers or inhibitors within 14 days of study entry. Substances in these categories include macrolide antibiotics (e.g. erythromycin, clarithromycin), azole antifungals (e.g. ketoconazole, fluconazole, itraconazole), rifampin, rifabutin, and phenytoin.
* Treatment with any investigational drug within 30 days of the first dose of study medication, and any neoplastic agent or radiotherapy other than local skin radiotherapy treatment within 12 weeks before starting study medication.
* Malabsorption, severe chronic diarrhoea or unable to maintain adequate oral intake.
* Treatment for an active infection (secondary to HIV-1).
* Hepatic insufficiency due to cirrhosis.
* Renal insufficiency.
* Excessive alcohol intake.
* Treatment with ritonavir.
* Treatment with protease inhibitors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2002-04; Primary Completion 2003-10 (Actual); Study Completion 2003-10

PRIMARY OUTCOMES:
Clearance of methadone at steady state in the presence and absence of nevirapine.

SECONDARY OUTCOMES:
Pharmacokinetics of methadone at steady state in the presence and absence of nevirapine

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BIL UK / Ireland
Locations (1):
- Department of Genito Urinary Medicine, St James' Hospital, Dublin, Ireland